CLINICAL TRIAL: NCT01009762
Title: Immunization With HIV-1 Peptides in Adjuvant for Treatment of Patients With
Brief Title: Immunization With HIV-1 Peptides in Adjuvant for Treatment of Patients With Chronic HIV-infection
Acronym: HIV-VAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gitte Kronborg (Other)
Collaborators: Statens Serum Institut (Other); Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other); Ministry of the Interior and Health, Denmark (Other Government)
Responsible Party: Sponsor-Investigator, Gitte Kronborg, Chief Medical Doctor, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT 2008-002980-15; 2008-002980-15 (EudraCT Number)
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: HIV INFECTIONS
Keywords: VACCINE; THERAPY; CELLULAR IMMUNITY; IMMUNITY
MeSH Terms: conditions — HIV Infections | interventions — Protein Subunit Vaccines; Peptides

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator): Sterile saline for injection is used as placebo arm. It is administered i.m. in the same way as for the active vaccine, week 0, 2, 4, 8.
- AFO-18 vaccine (Active Comparator): the intervention is injection of the experimental therapeutic peptide vaccine (AFO-18) consisting of 18 peptides in CAF01 adjuvant intra muscularly (i.m.) week 0, 2, 4, 8
  Interventions: Biological: peptide vaccine (AFO-18)

INTERVENTIONS:
Biological: peptide vaccine (AFO-18) — 18 Peptides (250 ug of each peptide) in Adjuvant CAF01 (= 625/125 ug DDA/TDB), i.m. injection week 0, 2, 4, 8.
  Other Names: DDA/TDB; peptides
  Arms: AFO-18 vaccine

SUMMARY:
Treatment: Immunization with a peptide-mix of 17 Clusters of Differentiation number 8 (CD8) T cell minimal epitopes and 3 Clusters of Differentiation number 4 (CD4) T cell epitopes and a new adjuvant (CAF01). The vaccine should induce cellular immunity against human immuno-deficiency virus type-1 (HIV-1).

Target group: Untreated healthy individuals with chronic HIV-1 infection who are not in antiretroviral treatment.

Purpose: The primary purpose is to evaluate tolerability and safety of the vaccine.

The secondary purpose is to evaluate the clinical effect of the vaccination treatment as measured by induction of new T cell immunity, lowering of HIV-1 ribonucleic acid (RNA) viral load in plasma, and improvement in the patient CD4 lymphocyte blood counts.

Design: The experiment is designed as a single-blinded, placebo-controlled phase 1 clinical trial in HIV-1 infected individuals in Denmark.

Numbers of individuals: 20 fully evaluable HIV-1-infected patients should enter the study (15 vaccine treated and 5 placebo(saline) treated controls).

The hypothesis is that a redirection of cytotoxic T lymphocyte (CTL) immunity to selected relatively immune silent (subdominant) but conserved CTL targets on multiple sites in HIV-1 could provide a better immune control of the virus replication. This could result in lowering of viral load thereby prolonging the time to antiretroviral therapy.

DETAILED DESCRIPTION:
The HIV-1 vaccine in this trial is designed to prevent disease in healthy already HIV-1 infected individuals not in anti-retroviral treatment by inducing a strong cellular immune response against several immune subdominant selected target points in the patient's HIV-1 virus. The vaccine treatment is not harmful but could potentially lower viral load and thus delay the time to acquired immuno deficiency syndrome (AIDS) disease or to the need of antiviral medicine and thereby limit the spread of HIV-1 in the population.

The patient's cellular immune response can only partly control the HIV-1 infection and eventually leads to a destruction of the immune system, opportunistic infections, and ultimately death. Normally the natural HIV-1 infection does not provide adequate immunity and vaccines must therefore induce a more potent and broader and more rationally directed immunity. Individuals that have this kind of strong immunity have lower viral-load and live longer. The vaccine in this study is designed to develop this kind of potent cellular immunity against HIV-1, so the virus is controlled better by the individual and spread in the population is limited.

This vaccine is designed to match most individual's cellular immune system (HLA tissue types) and several conserved target points in the individual's own HIV-1 virus. On the basis of our previous vaccine trial of HIV vaccination of HIV-infected individuals in Denmark and years of research, we have been able to develop this HIV-1 vaccine. Our vaccine contains 18 peptides (15 major histocompatibility complex class 1 (MHC-I) restricted CD8-t-cell epitopes and 3 MHC class-II restricted CD4 T-cell epitopes) in a mix and should induce cellular immune responses to several conserved target points identified in HIV-1. Our vaccine is composed of 18 peptides in a lipid based adjuvant Cationic Adjuvant Formulation number 1 (CAF01) composed of dimethyl-deoctadecylammonium (DDA) and trehalose-dibehenate (TDB) and is deemed safe and the technique is simple and also called 'peptide vaccination'. This and similar techniques have been tried in several studies against virus diseases around the world.

We want to know to which degree it is possible to immunize already HIV¬ 1 infected individuals to prolong the healthy period and prevent disease before initiation of antiviral medicine or other treatments of AIDS. In the present immunization study, healthy HIV-1 infected individuals not in treatment in Denmark will be invited to participate. This vaccine study will examine the immune responses and effects of the vaccine on these healthy HIV-1-infected individuals. The first purpose is first to determine if there are any side-effects of the vaccine. From several trials on animals and humans and in our own recent HIV vaccination trial on HIV-1 infected individuals in Denmark, with very similar vaccine techniques (peptides in autologous Dendritic Cells (DC) no serious side-effects has been observed. The second purpose is to examine if the vaccine induces the expected immune responses in HIV-1 infected individuals and how it enforces and supplements the already existing 'own' immune response of the infected individual. Finally, a clinical beneficial effect (on viral load and CD4 counts) of our vaccine will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 seropositive with measurable viral load >10e3 copies/ml and CD4+ T-cell count >400 CD4+ cells/µl
* Not in Antiretroviral Therapy (>1 year)
* Male or female with age between 18 and 60 years, where females are not breastfeeding, are not pregnant and use contraception until at least 3 months after end of vaccinations
* Normal values for the area of liver and kidney enzymes, blood cell count with differential counts e.g. white blood cells, lymphocytes, platelets, thrombocytes, and Hemoglobin
* Expected to follow the instructions
* Written informed consent after oral and written information

Exclusion criteria:

* Vaccinated with other experimental vaccines within 3 months before the first vaccination
* Treated with immune modulating medicine within 3 month before the first immunization
* Other significant active chronic infectious diseases likely to influence the HIV-1 infection, like Hepatitis B Virus (HBV), Hepatitis C Virus (HCV)
* Significant medical disease as judged by the investigators, for example severe asthma/chronic obstructive lung disease (COLD), badly regulated heart disease, insulin-dependent diabetes mellitus
* Severe allergy or earlier anaphylactic reactions
* Active autoimmune diseases
* Simultaneous treatment with other experimental drugs
* Laboratory parameters outside the 'normal' range for the area and which are considered clinically significant
* Pregnancy and/or brest feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Kronborg, MD, Principal Investigator — Hvidovre University Hospital; Anders Fomsgaard, MD, Study Director — Statens Serum Institut; Jan Gerstoft, MD, Study Chair — University of Copenhagen
Locations (1):
- Department Infectious Diseases, Hvidovre university hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Kloverpris H, Karlsson I, Bonde J, Thorn M, Vinner L, Pedersen AE, Hentze JL, Andresen BS, Svane IM, Gerstoft J, Kronborg G, Fomsgaard A. Induction of novel CD8+ T-cell responses during chronic untreated HIV-1 infection by immunization with subdominant cytotoxic T-lymphocyte epitopes. AIDS. 2009 Jul 17;23(11):1329-40. doi: 10.1097/QAD.0b013e32832d9b00. PMID 19528789
- [Derived] Karlsson I, Brandt L, Vinner L, Kromann I, Andreasen LV, Andersen P, Gerstoft J, Kronborg G, Fomsgaard A. Adjuvanted HLA-supertype restricted subdominant peptides induce new T-cell immunity during untreated HIV-1-infection. Clin Immunol. 2013 Feb;146(2):120-30. doi: 10.1016/j.clim.2012.12.005. Epub 2012 Dec 21. PMID 23314272

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the infectious disease department at the University hospitals
Pre-assignment Details: 20 participant numbers were randomised to vaccine or placebo but at the deadline for expiring of the vaccine only 11 participants were enrolled but all 11 completed the study
Groups:
- AFO-18 Vaccinated: Patients receiving the experimental therapeutic vaccine
Period: Overall Study
Arm/Group | Saline | AFO-18 Vaccinated
Started | 1 | 10
Primary Outcome | 0 (no Serious Adverse Events (SAE), no treatment related side effects DLT grade 3 or more) | 0 (no SAE, no treatment related side effects DLT grade 3 or more)
Completed | 1 (according to randomization this one participant received placebo) | 10 (10 participants received vaccine)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | AFO-18 Vaccinated | Total
Number analyzed (Participants) | 1 | 10 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 10 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 10 | 11
Region of Enrollment [Number; unit: participants]
  Denmark | 1 | 10 | 11
Clusters of Differentiation 4 (CD4) T-cells >400 cells/mm^3 [Number; unit: participants] | 1 | 10 | 11
Absence of T cell reaction to all vaccine peptides [Number; unit: participants] | 1 | 10 | 11
Viral load >10^3/mm^3 plasma [Number; unit: participants] — Numbers of participants with Viral Load in plasma above 1000 copies per ml
  participants | 1 | 10 | 11

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Treatment Related Side Effects (DLT = Reaction 3 or More)
Description: the numbers of treatment related side effects (DLT = reaction 3 or more) are registered for participants
Time Frame: up to 6 months after end of treatment
Population: Interview, questionaire, objective examination by medical doctor, blood testing for hematology, clinical chemistry, CD4 counts, HIV-1 viral load
Measure: Number; unit: side effects
Groups:
- Vaccinee: participants receiving the vaccine
- Placebo: participants receiving placebo (=saline)
Arm/Group | Vaccinee | Placebo
Number analyzed (Participants) | 10 | 1
side effects | 0 | 0

2. Secondary Outcome: Number of Participants With New T Cell Response to the Vaccine Target Epitopes
Description: Number of Participants with New T Cell Response to the Vaccine Target Epitopes as Measured by Intracellular Cytokine Stain Flowcytometry (IC-FACS) and/or IFNg-ELISPOT Analysis.
  Criteria's for meeting anticipated secondary end-point was that >50% of vaccinees reacted with new Clusters of differentiation 8 (CD8) T-cell and/or Clusters of differentiation 4 (CD4) T-cell response to al least one of the vaccine target epitopes as measured by IC-Facs and/or interferon-gamma (IFNg) - Enzyme-Linked ImmunoSpot (ELISPOT) assays.
Time Frame: 10-14 days or 3 months or 6 months after last immunisation
Population: Peripheral Blood Mononuclear Cells (PBMC) from blood was measured in IFNg-ELISPOT and/or Intracellular Cytokines (ICS) Flowcytometry for T cell responses. All 10 vaccinee developed a new T cell immune response to at least one vaccine epitope. The saline placebo did not develop any new t cell responses.
Measure: Number; unit: participants
Arm/Group | Saline | AFO-18 Vaccinated
Number analyzed (Participants) | 1 | 10
participants | 0 | 10

3. Secondary Outcome: Numbers of Participants With Lowering of HIV RNA Viral-load
Description: HIV-1 RNA Viral load was measured by Quantitative-PCR in plasma as numbers of virus RNA copies/mm^3 relative to baseline viral-load for each participant. The numbers of participant with lowering of HIV RNA plasma Viral-load is counted at base-line and at 6 months (end of study) and provided in the table (analysis population description) and the number of participants that showed lowering of viral-load was counted.
  Criteria for this anticipated end-point was a significant lowering of HIV RNA viral-load in >50% of responders (defined as participants with new T-cell responses).
Time Frame: up to 6 months after treatment stop
Population: the numbers of participants that showed changes (lowering of) in Viral load (measured as HIV-1 RNA copies/mm^3 plasma in commercial quantitative PCR) at end of study (6 months after vaccination) relative to base-line viral-load was counted at 6 month after vaccination (end of study)
Measure: Number; unit: participants
Arm/Group | Saline | AFO-18 Vaccinated
Number analyzed (Participants) | 1 | 10
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Vaccinee: participants receiving the vaccine called "AFO-18"
- Placebo: Participants receiving placebo (saline)
Arm/Group | Vaccinee | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/1
Other Adverse Events (participants affected / at risk) | 0/10 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No